CLINICAL TRIAL: NCT01220323
Title: Transcranial Direct Current Stimulation for Chronic Pain Relief
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Silviu Brill MD, Tel aviv Sourasky medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-10-SB-396-CTIL
Record Dates: First submitted 2010-10-06; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Chrronic Pain Patients
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- direct current stimulation (Active Comparator): The participants will be divided to 2 groups of 50 each. One group will receive 5 days period of 20 min 2mA tDCS over the lt M1 and the other will receive sham stimulation. X week later the groups will switch to the other arm.
  Interventions: Device: direct current stimulation
- sham stimulation (Sham Comparator)
  Interventions: Device: direct current stimulation

INTERVENTIONS:
Device: direct current stimulation — Patients will receive sham tDCS or real tDCS in a 5-day period of treatment in a randomized, sham controlled study. The participants will be divided to 2 groups of 50 each. One group will receive 5 days period of 20 min 2mA tDCS over the lt M1 and the other will receive sham stimulation. X week later the groups will switch to the other arm
  Arms: direct current stimulation
Device: direct current stimulation — Patients will receive sham tDCS or real tDCS in a 5-day period of treatment in a randomized, sham controlled study. The participants will be divided to 2 groups of 50 each. One group will receive 5 days period of 20 min 2mA tDCS over the lt M1 and the other will receive sham stimulation. X week later the groups will switch to the other arm
  Arms: sham stimulation

SUMMARY:
In the present study, the investigators intend to investigate whether anodal transcranial direct current stimulation (tDCS) may be effective in reducing pain in chronic pain patients.

DETAILED DESCRIPTION:
tDCS is a noninvasive brain stimulation technique that utilizes low amplitude direct currents applied via scalp electrodes to modulate the level of cortical excitability.Several studies have demonstrated that tDCS applied over the sensory-motor cortex has been able to decrease pain sensation and to increase pain threshold in healthy subjects and in chronic pain patients.

The aim of this study was to test whether daily sessions of anodal tDCS repeated for 5 consecutive days may be effective in reducing pain in a large number of chronic pain patients.

Patients will receive sham tDCS or real tDCS in a 5-day period of treatment in a randomized, sham controlled study. The participants will be divided to 2 groups of 50 each. One group will receive 5 days period of 20 min 2mA tDCS over the lt M1 and the other will receive sham stimulation. X week later the groups will switch to the other arm.

Pain will be measured using visual analog scale (VAS) for pain and the short form McGill questionnaire (SF-MPQ). Disability will be measured using the ( Pain Disability Index (PDI) of Life-54 scale (MSQoL-54). Depressive symptoms and anxiety will also be evaluated using the Center for Epidemiological Studies-Depression Scale and the State-trait Anxiety Inventory (STAI). Cognitive function will be mesured using minimental test. Evaluations will be performed at baseline, immediately after the end of treatment, and once a week during a 3-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* chronic pain patients VAS > 4

Exclusion Criteria:

* pregnancy
* scalp lacerations
* History of seizures
* metal implants in the head
* heart pace maker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 5 days

SECONDARY OUTCOMES:
Avaluation of tDCS treatment for chronic pain on disability, depression, anxiety, and cognition of treated patients. | 5 days